CLINICAL TRIAL: NCT07136987
Title: A Randomized Controlled Trial of 2 Disease-Modifying Drugs (Metformin and N-acetylcysteine ) to Promote TB Lung Function Recovery (TB-MET-NAC)
Brief Title: A Trial of 2 Disease-Modifying Drugs (Metformin and N-acetylcysteine ) to Promote TB Lung Function Recovery
Acronym: TB-MET-NAC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Open Source Pharma Foundation (Other)
Collaborators: National Institute for Research in Tuberculosis, Chennai, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUR1-22-465 TB-MET-NAC
Record Dates: First submitted 2025-08-05; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Tuberculosis
Keywords: lung function; FEV1; relapse
MeSH Terms: conditions — Tuberculosis; Recurrence | interventions — Metformin; Acetylcysteine; Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1:1 to the 3 arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metformin plus SOC (Experimental): Metformin 1500 mg total daily for 6 months plus standard TB treatment
  Interventions: Drug: Metformin
- N-acetylcysteine (NAC) plus SOC (Experimental): NAC 3600 mg total daily for 6 months plus standard TB treatment
  Interventions: Dietary Supplement: N-Acetylcysteine (NAC) Treatment
- Control (SOC) (Active Comparator): Standard TB treatment alone
  Interventions: Combination Product: Standard TB treatment

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg QAM x 1 wk, then 500 mg BID x 1 wk, then 1000 mg QAM and 500 mg QPM, plus standard TB treatment
  Arms: Metformin plus SOC
Dietary Supplement: N-Acetylcysteine (NAC) Treatment — N-acetylcysteine (NAC) 1800 mg orally twice daily plus standard TB treatment
  Arms: N-acetylcysteine (NAC) plus SOC
Combination Product: Standard TB treatment — Standard TB treatment
  Arms: Control (SOC)

SUMMARY:
Tuberculosis is a leading global cause of morbidity and mortality. Even if cured, a majority patients are left with bronchiectasis and fibrosis, permanent conditions that impair lung function. Large cohort studies have confirmed that even modest loss of lung function is associated with excess mortality risk. This study will examine if two treatments, metformin and N-acetylcysteine (NAC), can promote the recovery of lung function in TB if given together with standard TB treatment. There currently are no drugs approved for this indication.

DETAILED DESCRIPTION:
Tuberculosis is a leading global cause of morbidity and mortality. Current treatments are inadequate, requiring patients closely adhere to multi-drug regimens that are long, complex, and often poorly tolerated and/or ineffective. Even if cured, a majority patients are left with bronchiectasis and fibrosis, permanent conditions that impair lung function, particularly causing loss of FEV1% (the maximal 1-second exhaled volume in relation to age, sex, and height). FEV1 loss has profound long-term health consequences. Large cohort studies have confirmed that even modest loss of FEV1, remaining within 'normal' limits, is associated with excess mortality risk. This is most pronounced in low-income countries where TB is most prevalent. This study will examine if two treatments, metformin and N-acetylcysteine (NAC), can promote the recovery of lung function in TB. There currently are no drugs approved for this indication.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed written consent (or, in the case of illiteracy, witnessed oral consent plus patient thumbprint) prior to undertaking any trial-related procedures.
* Body weight (in light clothing without shoes) between 30 and 90 kg.
* Radiographic evidence of pulmonary tuberculosis
* Positive Xpert TB/RIF (original or Ultra) for MTB
* RIF susceptibility diagnosed by Xpert TB/RIF, with subsequent culture confirmation
* FEV1≤65% of predicted
* Eligible for treatment with a 6-month regimen comprised of INH, RIF, EMB, and PZA
* If sexually active, willing to use effective contraceptive methods for a period of 9 months (3 months post-study treatment)
* HIV-1 seronegative, or if HIV-1 seropositive, presenting to a non-India clinical site with a CD4 T cell count ≥100/µl and either receiving ART or willing to start ART during study participation
* SARS-CoV-2 PCR or antigen test negative, or if positive, either fully vaccinated against Covid-19 or with D-dimer <1 µg/ml
* eGFR ≥30 ml/min/1.73 m2 (CKD EPI 2009)

Exclusion Criteria:

* Any condition for which participation in the trial, as judged by the investigator, could compromise the well-being of the subject or prevent, limit or confound protocol specified assessments
* Currently pregnant or nursing, or pregnancy planned in next 12 months
* Is critically ill, and in the judgment of the investigator has a diagnosis likely to result in death during the trial or the follow-up period.
* TB meningitis or spondylitis, or other forms of severe tuberculosis with high risk of a poor outcome as judged by the investigator.
* History of allergy or hypersensitivity to any of the trial therapies or related substances.
* History of a chronic lung condition (including COPD or asthma) requiring treatment in the previous year
* Having participated in other clinical trials with investigational agents within 8 weeks prior to trial start or currently enrolled in an investigational trial.
* Prior TB treatment in the preceding 6 months, other than within the 7 days immediately prior to enrollment.
* Angina pectoris requiring treatment with nitroglycerin or other nitrates
* Cardiac arrhythmia requiring medication, or any clinically significant ECG abnormality, in the opinion of the investigator
* History of diabetes mellitus requiring treatment with metformin or resulting in hospitalization for hyper- or hypoglycaemia within the past year prior to start of screening
* Use of systemic corticosteroids within the past 28 days.
* Patients requiring treatment with medications not compatible with rifampin, such as HIV-1 protease inhibitors
* History of Pneumoconiosis.
* Subjects with any of the following abnormal laboratory values: hemoglobin <8 g/dL, platelets <100x109 cells/L, serum potassium <3.5 mM/L, alanine aminotransferase (ALT) ≥2.0 x ULN, alkaline phosphatase (AP) >5.0 x ULN, total bilirubin >1.5 mg/dL, HbA1c >6.5 %

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1104 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
FEV1 | month 18
  FEV1 after adjustment for baseline covariates including FEV1, in a superiority comparison
Favourable treatment outcome | 18 months
  Proportion of participants achieving a favourable treatment outcome (other than death, failure, recurrence, loss, default) in a non-inferiority comparison

SECONDARY OUTCOMES:
Other measures of lung function | Through month 18
  Changes in FEV1 and FVC
Microbiology | Through month 6
  Clearance of MTB from sputum measured as time to stable culture conversion and as rate of change in time to detection of MTB in automated liquid cultures (MGIT TTP)
Pharmacology | After 1 month of TB treatment
  Plasma TB drug exposures (Cmax and AUC0-24) using population PK modeling
Serious and non-serious adverse events | Through month 18
  The numbers of serious and non-serious adverse events
Radiography | 18 months
  Proportion of patients with persisting lung cavities on chest X ray
Immunology | 2, 6, and 18 months
  Blood measurements of inflammation (CRP) and immune function (IFN)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wallis, MD, Principal Investigator — OSPF and Aurum Institute

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD will be shared after the publication of the primary trial manuscript.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available after the publication of the primary manuscript. The end date has not yet been determined.
Access Criteria: Qualified investigators.
URL: https://tbportals.niaid.nih.gov/

REFERENCES:
- [Background] Pavan Kumar N, Padmapriyadarsini C, Nancy A, Tamizhselvan M, Mohan A, Reddy D, Ganga Devi NP, Rathinam P, Jeyadeepa B, Shandil RK, Guleria R, Singh M, Babu S. Effect of Metformin on systemic chemokine responses during anti-tuberculosis chemotherapy. Tuberculosis (Edinb). 2024 Sep;148:102523. doi: 10.1016/j.tube.2024.102523. Epub 2024 Jun 1. PMID 38850838
- [Background] Kumar AKH, Kadam A, Karunaianantham R, Tamizhselvan M, Padmapriyadarsini C, Mohan A, Jeyadeepa B, Radhakrishnan A, Singh UB, Bapat S, Mane A, Kumar P, Mamulwar M, Bhavani PK, Haribabu H, Rath N, Guleria R, Khan AM, Menon J; METRIF Team. Effect of Metformin on Plasma Exposure of Rifampicin, Isoniazid, and Pyrazinamide in Patients on Treatment for Pulmonary Tuberculosis. Ther Drug Monit. 2024 Jun 1;46(3):370-375. doi: 10.1097/FTD.0000000000001149. Epub 2023 Nov 28. PMID 38019456
- [Background] Padmapriydarsini C, Mamulwar M, Mohan A, Shanmugam P, Gomathy NS, Mane A, Singh UB, Pavankumar N, Kadam A, Kumar H, Suresh C, Reddy D, Devi P, Ramesh PM, Sekar L, Jawahar S, Shandil RK, Singh M, Menon J, Guleria R. Randomized Trial of Metformin With Anti-Tuberculosis Drugs for Early Sputum Conversion in Adults With Pulmonary Tuberculosis. Clin Infect Dis. 2022 Aug 31;75(3):425-434. doi: 10.1093/cid/ciab964. PMID 34849651
- [Background] Mapamba DA, Sabi I, Lalashowi J, Sauli E, Buza J, Olomi W, Mtafya B, Kibona M, Bakuli A, Rachow A, Velen K, Hoelscher M, Ntinginya NE, Charalambous S, Churchyard G, Wallis RS; TB SEQUEL consortium. N-acetylcysteine modulates markers of oxidation, inflammation and infection in tuberculosis. J Infect. 2025 Feb;90(2):106379. doi: 10.1016/j.jinf.2024.106379. Epub 2025 Jan 3. PMID 39756697
- [Background] Wallis RS, Sabi I, Lalashowi J, Bakuli A, Mapamba D, Olomi W, Siyame E, Ngaraguza B, Chimbe O, Charalambous S, Rachow A, Ivanova O, Zurba L, Myombe B, Kunambi R, Hoelscher M, Ntinginya N, Churchyard G. Adjunctive N-Acetylcysteine and Lung Function in Pulmonary Tuberculosis. NEJM Evid. 2024 Sep;3(9):EVIDoa2300332. doi: 10.1056/EVIDoa2300332. Epub 2024 Aug 27. PMID 39189858